CLINICAL TRIAL: NCT02969538
Title: Effect of Shortening the Etching Time on the Clinical Performance of Resin Composite Restorations in Primary Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal de Santa Maria (Other)
Responsible Party: Principal Investigator, Tathiane Lenzi, Principal investigator, Universidade Federal de Santa Maria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UFSantaMaria1
Record Dates: First submitted 2016-04-04; First posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries | interventions — phosphoric acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Total etching time (Other): Dentin etching (35% phosphoric acid) by time recommend by manufacturer (15 seconds)
  Interventions: Other: Total etching time
- Half-reduced etching time (Experimental): Dentin etching (35% phosphoric acid) by 7 seconds
  Interventions: Other: Half-reduced etching time

INTERVENTIONS:
Other: Total etching time — Apply 35% phosphoric acid on dentin and enamel by 15 seconds.
  Other Names: (dental conditioner - 35% phosphoric acid)
  Arms: Total etching time
Other: Half-reduced etching time — Apply 35% phosphoric acid on enamel by 15 seconds and dentin by 7 seconds.
  Other Names: (dental conditioner - 35% phosphoric acid)
  Arms: Half-reduced etching time

SUMMARY:
The aim of this study is to evaluate the effect of shortening the etching time on the 18-month clinical performance of resin composite restorations in primary molars after partial carious removal. This randomized clinical trial will include subjects (5-10 year-old children) selected at Pediatric Clinic of Federal University of Santa Maria. The sample will consist of 70 primary molars presenting active cavitated carious lesions (with radiographic involvement of the outer half of the dentin), located on the occlusal surface. The sample will be randomly divided into two groups according to the etching time of the dentin prior adhesive application (Adper Single Bond 2; 3M ESPE): recommend by manufacturers (15 seconds) and half-reduced etching time (7 seconds). The restorations will be clinically followed every 6 months for up to 18-month using the FDI criteria for clinical evaluation. Survival estimates for restoration longevity will be evaluated using the Kaplan-Meier method.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of shortening the etching time on the 18-month clinical performance of resin composite restorations in primary molars after partial carious removal. This randomized clinical trial will include subjects (5-10 year-old children) selected at Pediatric Clinic of Federal University of Santa Maria. The sample will consist of 70 primary molars presenting active cavitated carious lesions (with radiographic involvement of the outer half of the dentin), located on the occlusal surface. The sample will be randomly divided into two groups according to the etching time of the dentin prior adhesive application (Adper Single Bond 2; 3M ESPE): applying of 35% phosphoric acid by 15 s - recommend by manufacturers and half-reduced etching time (7 s). The restorations will be clinically followed every 6 months for up to 18-month using the FDI criteria for clinical evaluation. Survival estimates for restoration longevity will be evaluated using the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

*Active carious lesion in middle dentin limited to the occlusal surfaces of primary molars.

Exclusion Criteria:

* Children who refuse or fail to cooperate with the completion of clinical procedure;
* Teeth without antagonist;
* Carious lesions in inner half of dentin;
* Presence of painful symptoms or signs of pulpal changes.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Failure of restorations | 18 months after restorations' placement

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Santa Maria, Santa Maria, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided